CLINICAL TRIAL: NCT03773172
Title: Study to Evaluate the Effects of Two Doses Over 48 Hours of MEDI6012 on Apolipoprotein B100 Metabolism in Subjects With Stable Atherosclerotic Cardiovascular Disease
Brief Title: Study to Evaluate the Effects of MEDI6012 on Apolipoprotein B100 Metabolism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to COVID-19
Sponsor: Columbia University (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Henry N. Ginsberg, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAS0459
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
Keywords: Lipid and Lipoprotein Metabolism
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Control Group (Placebo Comparator): Subjects will receive placebo treatment to mimic active treatment.
  Interventions: Drug: Placebo
- Active treatment (Active Comparator): IV push loading dose of 300 mg MEDI6012 followed by a 150 mg maintenance dose of MEDI6012 at 48 hours.
  Interventions: Drug: MEDI6012

INTERVENTIONS:
Drug: MEDI6012 — MEDI6012 is recombinant human lecithin-cholesterol acyltransferase (rhLCAT), an approximately 60 kilodalton, glycosylated, single-chain protein consisting of 416 amino acids produced via Chinese hamster ovary cell culture. It is being explored as an acute treatment to reduce the risk of recurrent cardiovascular events as an adjunct to the standard of care in patients with acute myocardial infarction (MI). MEDI6012 and ACP501 have the identical amino acid sequence and are therefore considered the same molecular entity.
  Other Names: Stable Isotopes
  Arms: Active treatment
Drug: Placebo — The placebo will mimic the active treatment.
  Other Names: Placebo compound provided by funding agency
  Arms: Placebo Control Group

SUMMARY:
This is a Phase 2, single-center, placebo controlled, double-blind, randomized crossover study to determine the effects of MEDI6012 on the metabolism of apolipoprotein B100 (apoB100) lipoproteins in individuals with stable atherosclerotic cardiovascular disease (ASCVD).

DETAILED DESCRIPTION:
Atherosclerosis, characterized by excess fat deposit in arteries, is a progressive and life-threatening condition. Therefore, treatments that can remove fat deposits from the arteries are being developed. These treatments may prevent subsequent heart attacks or other cardiovascular events, addressing an unmet medical need. MEDI16012 is a new drug that targets a substance produced by the body to assist participants in breaking down the bodies "good" fat. The investigators are interested in understanding why MEDI6012 increases the good fat, but also why it increases other types of "bad" fat such as low-density lipoprotein-C (LDL-C).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects (non-childbearing potential for females) ages 35 through 80 years at the time of screening who are capable of providing informed consent prior to screening and any protocol-related procedures.
2. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act (HIPAA) in the USA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. Ability to complete and meet all eligibility requirements for randomization within 28 days of informed consent (56 days if washing out from lipid altering agent other than statins or ezetimibe).
4. A diagnosis of stable atherosclerotic cardiovascular disease (CVD) documented prior to screening:

   * Coronary artery disease defined as a history of prior myocardial infarction, coronary revascularization, history of coronary atherosclerosis based on invasive or non-invasive imaging, and/or abnormal stress testing diagnostic of coronary artery disease.
   * Carotid artery disease (extracranial internal carotid artery (ICA) stenosis) defined as evidence of carotid atherosclerosis by carotid imaging, or history of percutaneous or surgical carotid revascularization
   * Peripheral artery disease defined as ankle-brachial index < 0.90 and claudication, or prior peripheral revascularization for ischemia, or evidence of lower extremity (below the inguinal ligament) atherosclerosis on invasive or noninvasive imaging
5. Currently receiving statin as standard of care, at a stable dose for ≥ 8 weeks prior to screening and intended to remain at a stable dose throughout the study duration. Subjects may also be receiving ezetimibe, 10 mg/day for ≥ 8 weeks prior to screening.
6. Nonsterilized males who are sexually active with a female partner of childbearing potential must use condom and spermicide from Day 1 through the end of their participation in the study. Because male condom and spermicide is not a highly effective contraception method it is strongly recommended that female partners of a male study subjects also use a highly effective method of contraception throughout this period.

Exclusion Criteria:

1. Unstable cardiovascular conditions within 3 months prior to screening, including acute coronary syndrome (ACS), stroke or transient ischemia attack, critical limb ischemia, non-elective arterial revascularization, life-threatening arrhythmias, or heart failure hospitalization.
2. Elective arterial revascularization (in any vascular territory) in the past 1 month. Any planned arterial revascularization (coronary, peripheral or carotid).
3. New York Heart Association (NYHA) Class III or IV congestive heart failure or treatment with advanced therapies (cardiac transplant, ventricular assist device, cardiac resynchronization therapy,and/or chronic IV inotropic support), or severe valvular heart disease.
4. Body mass index < 18 or > 45.
5. Lipid measurements with any of the following:

   1. Triglycerides (TG) > 400 mg/dL
   2. LDL-C > 120 mg/dL
   3. High-density lipoprotein C (HDL-C) > 70 mg/dL for males or > 80 mg/dL for females.
6. Clinically significant vital sign abnormalities at screening or on Day -1:

   1. Systolic blood pressure (BP) < 90 or >160 mm Hg
   2. Diastolic BP > 100 mm Hg
7. Females currently breastfeeding or of childbearing potential. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are not postmenopausal; defined as 12 months with no menses without an alternative medical cause and a follicle-stimulating hormone level in the central laboratory's normal range for post-menopausal phase is required at screening.
8. Use of lipid-lowering medications, with the exception of statins and ezetimibe, and the following dietary supplements: ≥ 2 grams/day of fish oil (≥ 2 grams/day docosahexaenoic acid (DHA) and EPA combined), ≥ 30 grams/day of flaxseed oil or ground flaxseed, red yeast extract, > 100 mg/day of niacin. At the investigator's discretion, subjects may undergo a 6-week washout period of any exclusionary lipid-lowering agents with the expectation that post-washout lipid levels will be rechecked and acceptable per above criteria.
9. History of any of the following:

   * Documented familial hypercholesterolemia
   * Chronic kidney disease defined by estimated glomerular filtration rate < 30 mL/min/1.73 m2 by the modification of diet in renal disease equation, or end stage renal disease treated with kidney transplant or renal replacement therapy
   * History of clinically overt chronic liver disease or biochemical evidence of liver disease
   * Poorly controlled endocrine disorder including:

     * Type 1 Diabetes excluded
     * Type 2 Diabetes Mellitus with glycated hemoglobin (HbA1c) > 8.0% as assessed at screening or
   * Uncontrolled thyroid disorder defined as thyroid stimulating hormone (TSH)> upper limit of normal (ULN) and abnormal free T4; subjects with thyroid deficiency should have received a stable dose of thyroid hormone for > 6 weeks prior to screening and have a normal TSH.
   * Current or previous use of systemic corticosteroids within 28 days prior to screening. Topical, intra-articular, intranasal, inhaled, and ophthalmic steroid therapies are allowed
   * History of severe infection or ongoing febrile illness within 30 days of screening, or a medical history of a chronic viral illness including hepatitis B or C virus, or human immunodeficiency virus (HIV).
   * History of active malignancy within 5 years (subjects with non-melanotic skin cancer may be included)
   * Any other disease or condition or laboratory value that, in the opinion of the investigator or medical monitor, would place the subject at an unacceptable risk or interfere with the evaluation of the investigative product.
   * Known allergy/hypersensitivity to any component of the investigational product formulation, other biologics, IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
10. Subjects who are legally institutionalized
11. Previous Exposure to rhLCAT
12. Concurrent enrollment in another clinical study of any investigational drug therapy or use of any biologicals within 6 months prior to screening or within 5 half-lives of an investigational agent or biologic, whichever is longer.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were enrolled; 2 participants withdrew consent prior to randomization and therefore were not included in the Participant Flow.
Groups:
- MEDI6012 First, Then Placebo: Participants will receive IV push loading dose of 300 mg MEDI6012on Day 0. On Day 2 (exactly 48 hours from Day 0 administration), they will receive the 2nd dose of 300 mg MEDI6012. After a 6-8 washout period, the participants will repeat the same protocol but will receive the placebo.
- Placebo, Then MEDI6012: Participants will receive IV push loading dose of 300 mg placebo on Day 0. On Day 2 (exactly 48 hours from Day 0 administration), they will receive the 2nd dose of 300 mg placebo. After a 6-8 washout period, the participants will repeat the same protocol but will receive MEDI6012.
Period: First Intervention (3 Days)
Arm/Group | MEDI6012 First, Then Placebo | Placebo, Then MEDI6012
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Washout (6 to 8 Weeks)
Arm/Group | MEDI6012 First, Then Placebo | Placebo, Then MEDI6012
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Second Intervention (3 Days)
Arm/Group | MEDI6012 First, Then Placebo | Placebo, Then MEDI6012
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected per Arm, thus cannot be presented per Arm.
Groups:
- Placebo Control or Active Treatment: Subjects will receive placebo treatment to mimic active treatment. Placebo: The placebo will mimic the active treatment.
  OR
  IV push loading dose of 300 mg MEDI6012 followed by a 150 mg maintenance dose of MEDI6012 at 48 hours.
  MEDI6012: MEDI6012 is recombinant human lecithin-cholesterol acyltransferase (rhLCAT), an approximately 60 kilodalton, glycosylated, single-chain protein consisting of 416 amino acids produced via Chinese hamster ovary cell culture. It is being explored as an acute treatment to reduce the risk of recurrent cardiovascular events as an adjunct to the standard of care in patients with acute myocardial infarction (MI). MEDI6012 and ACP501 have the identical amino acid sequence and are therefore considered the same molecular entity.
  (Study is double-blind)
Arm/Group | Placebo Control or Active Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Fractional Clearance Rate (FCR) of Lipoprotein B (Pools/Day)
Description: FCR is the rate of synthesis and clearance of soluble lipoprotein B in participants per day.
Time Frame: Up to 48 hours from first dose
Measure: Mean (Standard Deviation); unit: pools/day
Groups:
- MEDI6012: Participants will receive IV push loading dose of 300 mg MEDI6012on Day 0. On Day 2 (exactly 48 hours from Day 0 administration), they will receive the 2nd dose of 300 mg MEDI6012.
- Placebo: Participants will receive IV push loading dose of 300 mg placebo on Day 0. On Day 2 (exactly 48 hours from Day 0 administration), they will receive the 2nd dose of 300 mg placebo.
Arm/Group | MEDI6012 | Placebo
Number analyzed (Participants) | 5 | 5
pools/day | 14.0 (6.0) | 10.0 (5.5)

2. Secondary Outcome: Production Rate (PR) of Apolipoprotein B100 (mg/kg/Day)
Description: Amount of Apolipoprotein B100 (measured as mg/kg) produced in participants per day.
Time Frame: Up to 48 hours from first dose
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | MEDI6012 | Placebo
Number analyzed (Participants) | 5 | 5
mg/kg/day | 14.2 (11.3) | 15.7 (3.2)

3. Other Pre Specified Outcome: ADA Measurement
Description: To access the immunogenicity of MEDI6012, anti-drug antibodies (ADA) will be measured.
Time Frame: Up to 60 days post administration of first dose
Population: Double-blind study terminated early due to COVID-19. Data was not collected for this outcome measure and therefore cannot be analyzed.
Arm/Group | MEDI6012 First, Then Placebo | Placebo, Then MEDI6012
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 60 days post administration of first dose.
Description: Data for Adverse Events were collected agnostic to the intervention.
Arm/Group | MEDI6012 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MEDI6012 (N=5) | Placebo (N=5)
Headache (General disorders) | 0 | 1
Blurry vision (Eye disorders) | 0 | 1
Insomnia (General disorders) | 0 | 1
Dyspnea (General disorders) | 0 | 1
Flushing (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Double-blind study was terminated early due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03773172/Prot_SAP_000.pdf